CLINICAL TRIAL: NCT07164144
Title: SAVE: School Ambassadors for Vaccine Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cynthia Rand, Professor, Pediatrics & Division Chief, General Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00010895
Record Dates: First submitted 2025-08-27; First posted 2025-09-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Immunization; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Vaccine Communication Training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Vaccine Communication Training — School personnel receive vaccine communication training + promotional materials
  Arms: Intervention

SUMMARY:
Influenza is associated with millions of cases of school absenteeism due to illness, hundreds of hospitalizations and thousands of deaths in the U.S. each year, which can be greatly reduced with influenza vaccination.

The goal of this randomized controlled trial is to learn if training school personnel in vaccine communication techniques and equipping schools with vaccine promotional materials targeting students and their parents/guardians increases the influenza vaccination rates of the student population within participating schools.

The main question it aims to answer is:

-Will flu vaccination rates be higher in intervention schools compared to control schools by the end of the intervention period?

Participating schools will:

* Have select school personnel (school nurses, coaches, teachers, etc.) complete an online training module and optional training workshop focused on vaccine communication [intervention arm only]
* Utilize vaccine promotional materials (posters, flyers, digital files for social media, etc.) provided by the study team during flu season [intervention arm only]
* Track student vaccination rates [intervention + control arm]

ELIGIBILITY:
Inclusion Criteria:

* A student enrolled in a participating school (intervention or control) for at least one year

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Flu vaccination rate | 8 months (one flu season August-March)

IPD SHARING:
Plan to Share IPD: No